CLINICAL TRIAL: NCT02138084
Title: Pharmacokinetic Interaction Study to Evaluate the Pharmacokinetic Effect of Rifabutin on BMS-626529, the Active Moiety of BMS-663068, With and Without Ritonavir in Healthy Subjects
Brief Title: Drug-drug Interaction (DDI) Rifabutin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 206282; AI438-041 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-05-13; First posted 2014-05-14 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Rifabutin; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: BMS-663068 + Rifabutin (Experimental): Regimen A: BMS-663068 tablet by mouth as specified
  Regimen B: BMS-663068 tablet with Rifabutin capsule by mouth as specified
  Interventions: Drug: BMS-663068; Drug: Rifabutin
- Cohort 2: BMS-663068 + Rifabutin + Ritonavir (Experimental): Regimen A: BMS-663068 tablet by mouth as specified
  Regimen C: BMS-663068 tablet, Rifabutin capsule and Ritonavir (RTV) capsule by mouth as specified
  Interventions: Drug: BMS-663068; Drug: Rifabutin; Drug: Ritonavir

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Drug: Rifabutin — Rifabutin
Drug: Ritonavir — Ritonavir
  Arms: Cohort 2: BMS-663068 + Rifabutin + Ritonavir

SUMMARY:
The purpose of this study is to provide dosing recommendations for the coadministration of BMS-663068 and Rifabutin with and without Ritonavir in upcoming Phase 3 studies and for prescribing information purposes

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

1. Signed Written Informed Consent

   a) Signed written informed consent must be obtained from the subjects in accordance with requirements of the study center's Institutional Review Board (IRB) or Independent Ethics Committee (IEC) before the initiation of any protocol-required procedures
2. Target Population

   * a) Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination findings, 12-lead ECG measurements, and clinical laboratory test results
   * b) Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive BMI = weight (kg)/[height (m)]2
   * c) Subject Reenrollment: This study permits the reenrollment of a subject that has discontinued the study as a pretreatment failure (ie, subject has not been randomized/has not been dosed). If reenrolled, the subject must be reconsented
3. Age and Reproductive Status

   * a) Men and women, ages 18 to 50 years, inclusive
   * b) Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study drug
   * c) Women must not be breastfeeding
   * d) WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of Rifabutin (13 days) plus 30 days (duration of ovulatory cycle) for a total of 43 days posttreatment completion
   * e) Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of Rifabutin (13 days) plus 90 days (duration of sperm turnover) for a total of 103 days posttreatment completion

Exclusion Criteria:

Medical History and Concurrent Diseases

* a) Any significant acute or chronic medical illness as determined by the Investigator.
* b) Current or recent (within 3 months of study drug administration) gastrointestinal disease
* c) Any major surgery within 4 weeks of study drug administration
* d) Any gastrointestinal surgery that could impact upon the absorption of study drug
* e) Intractable diarrhea (≥6 loose stools per day for at least 7 consecutive days) within 30 days prior to the first dose of study drug
* f) History of acute or chronic pancreatitis
* g) History of active or latent tuberculosis or any recent exposure to someone with tuberculosis
* h) History of uveitis and/or current eye or vision problems with the exception of corrective lenses
* i) Contact lens use during study drug administration or the need for contact lenses during study drug administration
* j) Donation of blood to a blood bank or in a clinical study (except screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma donation only)
* k) Blood transfusion within 4 weeks of study drug administration.
* l) History of any hemolytic disorders, including drug-induced hemolysis.
* m) Inability to tolerate oral medication
* n) Inability to be venipunctured and/or tolerate venous access
* o) Recent (within 6 months of study drug administration) history of smoking or current smokers
* p) Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV), Diagnostic Criteria for Drug and Alcohol Abuse
* q) Any other sound medical, psychiatric, and/or social reason as determined by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2014-07-24 (Actual); Study Completion 2014-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-626529 | Day 2 to Day 15
Area under the concentration-time curve in 1 dosing interval [AUC(TAU)] of BMS-626529 | Day 2 to Day 15

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) of BMS-626529 | Day 2 to Day 15
Concentration at 12 hours after dosing (C12) of BMS-626529 | Day 2 to Day 15
Trough observed plasma concentration (Ctrough) of BMS-626529 (predose) | Day 2 to Day 15
Safety and tolerability include incidence of adverse events (AEs), serious AEs (SAEs), AEs leading to discontinuation, deaths, marked laboratory abnormalities, and abnormalities in vital signs, physical examination, and 12-lead electrocardiograms (ECGs) | Up to Day 30 after discontinuation of dose (approximately 45 days)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States